CLINICAL TRIAL: NCT02817438
Title: Research on Anxiety and Depression: Computer-Assisted Therapy
Acronym: RADCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tali Manber Ball, PhD, Postdoctoral Scholar, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-36790
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Mood Disorders; Anxiety Disorders
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online Intervention (Experimental): Participants randomized to the online intervention arm will be given access to the Good Days Ahead program for 12 weeks.
  Interventions: Behavioral: Good Days Ahead
- Waitlist (No Intervention): Participants randomized to the waitlist arm will wait for 12 weeks without doing an online intervention.

INTERVENTIONS:
Behavioral: Good Days Ahead — Good Days Ahead is a web-based program based on the principles of Cognitive Behavioral Therapy (CBT). It can be used to supplement traditional psychotherapy, or as a stand-alone intervention. There are 9 lessons that address Thinking Skills, Behavioral Skills, Schemas, and Coping Tools. Lessons include videos from expert therapists and a Practice Section in which patients complete forms for self-monitoring symptoms and challenging negative thoughts.
  Arms: Online Intervention

SUMMARY:
This study examines how online self-guided programs can improve mood and anxiety symptoms. These programs use exercises from Cognitive-Behavioral Therapy, which is an evidence-based treatment for depression and anxiety. The purpose of this study is to learn who will do best with the online format. Our aim is to learn for whom online self-guided interventions are most efficacious. This knowledge is important because it will help inform clinicians and patients about who might benefit from this type of intervention versus who would need the assistance of a therapist. More specifically, we hope to figure out who would benefit from solely an online intervention and who would benefit from an online intervention in addition to other treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the RAD study in our laboratory

RAD study inclusion criteria are:

* 18+ years of age
* Fluent and literate in English
* Can provide informed consent
* fMRI scanning eligibility, including no evidence of any form of metal embedded in the body (e.g., metal wires, nuts, bolts, screws, plates, sutures)

Exclusion Criteria:

* Anyone who has not already completed the RAD study will be excluded.

RAD study exclusion criteria are:

* Presence of suicidal ideations representing imminent risk
* General medical condition, disease, or neurological disorder that interferes with the assessments
* Mild traumatic brain injury (history of physical brain injury or blow to the head resulting in loss of consciousness greater than five minutes) and which could interfere with doing the assessments
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with ability to complete the assessments
* Unable and/or unlikely to follow the study protocols
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-06; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Depression and Anxiety Composite Score | 12 weeks
  Composite score combining 3 measures of depression and/or anxiety (PHQ-9, BAI, DASS)

SECONDARY OUTCOMES:
Quality of Life | 12 weeks
  WHOQOL scale

CONTACTS AND LOCATIONS:
Overall Officials: Tali Ball, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States